CLINICAL TRIAL: NCT01381939
Title: Induction of Labor in Intrahepatic Cholestasis of Pregnancy
Acronym: ILICP
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Prof Hanns-Ulrich Marschall, Sahlgrenska Academy, University of Gothenburg
Other Study IDs: 6647416
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2010-03

CONDITIONS: Intrahepatic Cholestasis
Keywords: Intrahepatic Cholestasis of Pregnancy; Induction of labor; Pregnancy; Caesarian section; Pruritus; IUFD
MeSH Terms: conditions — Cholestasis, Intrahepatic; Intrahepatic Cholestasis of Pregnancy; Pruritus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Induction of labor in ICP: Induction of laborin women with ICP
- Induction of labor in women with no ICP: No ICP
- ICP and spontanius delivery

SUMMARY:
Induction of Labour in Intrahepatic Cholestasis of Pregnancy (ICP) has become a common procedure in management of ICP to avoid fetal complications. Surprisingly, this empirical approach has not been evaluated as to delivery complications and fetal outcome as yet. The investigators now examine weather ICP affects (i) delivery procedures chosen, in particular the incidence of caesarian section, (ii)fetal and maternal outcome in induced labor, and (iii)possible impact of bile acids and UDCA treatment in a retrospective cohort study based on approximately 5000 induced deliveries at Danderyd Hospital, Karolinska Institutet, Stockholm. The investigators analyze data on on previous deliveries, BMI, medical history and medical book data. Primary endpoint is the risk of caesarian section.

ELIGIBILITY:
Inclusion Criteria:

* ICP during pregnancy and induction of labor ICP and spontaneous delivery No ICP but induction of labor

Exclusion Criteria:

* No ICP spontaneous delivery
* Elective caesarian section

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Swedish women affected by ICP delivering at Danderyd Hospital between year 2000-2006.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2000-01; Primary Completion 2006-12 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Cesarean section | 32 to 40 weeks

SECONDARY OUTCOMES:
Bleeding | 32 to 40 weeks
Abruptio placentae | 32 to 40 weeks
APGAR | 32 to 40 weeks